CLINICAL TRIAL: NCT00740558
Title: Heart Rate Variability Modulation Following a Manipulation in Pain Free Patients Versus Patients in Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec a Montréal (Other)
Responsible Party: Dr Richard Roy DCMScPhD(c), UQAM
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 051934
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Last update posted 2008-08-27 (Estimated); Status verified 2008-08

CONDITIONS: Low Back Pain
Keywords: HRV; Activator; Chiropractic; VLF; HF; LF; LF/HF
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Two groups received a traditional chiropractic adjustment of the lumbar 5 and the other group received a manually assisted mechanical force adjustment of the lumbar 5.
  Interventions: Procedure: Activator methods technique; Procedure: Traditional chiropractic adjustment
- 2 (Sham Comparator): The investigators had two groups, one for each chiropractic technique used in the research project and we had a control group
  Interventions: Procedure: Activator methods technique; Procedure: Traditional chiropractic adjustment

INTERVENTIONS:
Procedure: Activator methods technique — Chiropractic adjustment by a manually assisted mechanical force
  Other Names: Activator methods
Procedure: Traditional chiropractic adjustment — Lumbar roll according to the Diversified technique of chiropractic adjusting
  Other Names: Lumbar roll

SUMMARY:
Background

The purpose of this study was to examine the heart rate variability (HRV) in the presence or the absence of pain in the lower back (L5), while receiving chiropractic care.

Methods

A total of 53 healthy participants were randomly assigned to a control, 2 treatment or 2 sham groups (n = 10 per group). Participants underwent an eight-minute acclimatizing period. The HRV tachygram (RR interval) data were recorded directly into a Suunto watch (model T6). The investigators analyzed the five minute pre-treatment and post treatments intervals. The spectral analysis of the tachygram was performed with the Kubios Software (University of Kuopio, Finland).

DETAILED DESCRIPTION:
Background The chiropractic profession has in the past utilized research results from other fields of and extrapolated them into their science and clinical interpretation 1-4. More recently, chiropractic researchers looked into autonomic nervous system (ANS) adaptations in an animal model following a mechanical stress to the spinal column 5, a noxious mechanical stimulation 6 or a spinal manipulation 7.

In the human model, several investigations have been done to measure modifications of the heart rate variability (HRV) following cervical 8 and thoracic manipulations 9 or in a multisite clinical study 10 where details of the manipulation site were not provided. The site of interest for the chiropractic intervention was defined at the level of the lumbar spine, left and right L-5. This site was selected because most studies 8-10 measuring HRV have used the cervical or thoracic component of the spine. The effect of the lumbar parasympathetic nervous system has not been evaluated. In these studies 8-10, changes were observed in various HRV variables, while in two of those studies 8, 9, where sham groups were included, the sham conditions did not demonstrate any changes in the reported HRV parameters. There are strong indications that HRV is a good marker of ANS activity 19-24. Thus, in the three above mentioned studies, it appears that chiropractic interventions have an effect on the ANS.

At present, however, no studies to evaluate whether a lumbar spinal manipulation would produce a change in the HRV have been reported. Thus, the present study seeks to measure the effect of a lumbar adjustment, with a manually assisted mechanical force, producing a chiropractic adjustment, in participants without lumbar pain and a traditional adjustment in participants with lumbar pain on HRV. The hypothesis being that a lumbar intervention would have an acute effect on the ANS as demonstrated by the modulation of HRV variables.

ELIGIBILITY:
Inclusion Criteria:

* Acute low back pain (pain group)
* Maintenance care for the pain free group and the control group

Exclusion Criteria:

* For the control group (pain)
* For the non pain group pain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2004-07; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Mean R-R interval, the number of pairs of adjacent NN intervals differing by more than 50 ms, and the proportion of NN intervals differing by more than 50 ms the very low frequency, the low frequency, the high frequency, the LF/HF ratio | Pre and post measurements of one intervention

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Roy, DCMScPhD(c), Principal Investigator — Université du Québec a Montréal
Locations (2):
- Canada (2):
  - Chiro-clinique Richard Roy, LaSalle, Quebec
  - Dr Richard Roy et Dr Fafard, LaSalle, Quebec